CLINICAL TRIAL: NCT06670391
Title: A Retrospective, Real-world, Electronic Medical Record-based Study on Patients With Liver Injury After the Administration of Novel Antineoplastic Agents
Brief Title: A Retrospective Study in Patients With Liver Injury After the Use of Novel Antineoplastic Agents
Status: Active, not recruiting | Type: Observational
Sponsor: Drug Induced Liver Disease Study Group (Other)
Responsible Party: Principal Investigator, Yimin Mao, Chairman, Drug Induced Liver Disease Study Group
Other Study IDs: GM_DILI_002
Record Dates: First submitted 2024-10-29; First posted 2024-11-01 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Liver Injury; Liver Injury, Drug-Induced
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is an open-enrollment, retrospective, observational study without interventions. Its primary objective is to understand 1) incidence of liver injury among all the hospitalized patient from participating centers after the administration of immune checkpoint inhibitors or molecularly targeted agents; 2) epidemiologic and clinical characteristics of liver injury, including suspected medications, clinical types, histological characteristics, severity, treatment and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Abnormality of liver biochemistry after the administration of any molecularly targeted agent or immune checkpoint inhibitor

Exclusion Criteria:

* Missing major baseline or clinical data
* Prior liver loco-regional therapy or surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All hospitalized patients from participating medical centers.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in ALT (alanine aminotransferase) | on day 10
  Absolute change

SECONDARY OUTCOMES:
Proportion of patients with normalized liver biochemistry | on day 3, 7, 10, 14, 21, and 30
  Count of subjects
Change in liver biochemistry | on day 3, 7, 10, 14, 21, and 30
  Absolute change
Time to normalization of liver biochemistry | up to 6 month
  Days
Proportion of patients with ≥ 50% reduction in liver biochemistry | on day 3, 7, 10, 14, 21, and 30
  Count of subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China